CLINICAL TRIAL: NCT01761032
Title: Dopamine Response to Ultraviolet Light in Frequent and Infrequent Tanners
Brief Title: Gauging Of Light Dependent Experiences Through Neuroimaging (GOLDEN)
Acronym: GOLDEN
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: STU 112011-012; R21AR063018 (NIH)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Compulsive and Infrequent Tanners
Keywords: Tanning; neuroimaging; dopamine; MRI; SPECT

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Infrequent tanners: Individuals who tan less than twice a week and do not meet modified DSM-IV criteria for tanning addiction.
  Interventions: Device: Tanning
- Compulsive Tanners: Individuals who tan more than 3 times per week in a tanning bed. Tanning must cause disruption in daily functioning. Must meet modified DSM-IV criteria for tanning addiction
  Interventions: Device: Tanning

INTERVENTIONS:
Device: Tanning — Participants will be placed under a tanning canopy for 4-10 minutes.

SUMMARY:
In the proposed study, the investigators will assess the brain's dopamine response to UVR light in individuals who use tanning beds both frequently and infrequently.

DETAILED DESCRIPTION:
UV radiation has recently been classified as a known human carcinogen by the US Department of Health and Human Services. Nevertheless, the voluntary exposure to sunlight continues unabated despite progressively increasing rates of ultraviolet radiation (UVR)-induced illness and death, particularly skin cancer. An increasingly common form of UVR administration is through the use of indoor tanning salons. Almost 30 million Americans, including 20% of 18-39 year olds, visit indoor tanning salons each year. Frequent and excessive tanning, despite a growing understanding by those who tan of the morbidity and mortality associated with tanning, suggests that UVR may impart rewarding effects beyond the assumed cosmetic benefits. Recent studies, in fact, have shown that up to 40% of both frequent beach and salon tanners exhibit signs and symptoms consistent with an addictive disorder, including an inability to decrease their tanning frequencies, compulsive tanning, and/or continued tanning despite adverse consequences. As the mesostriatal dopaminergic pathway plays a key role in reward and addiction, the investigators propose to extend this novel finding by directly assessing the mesostriatal dopaminergic reward pathway in compulsive and infrequent tanners. This pathway plays a key role in the experience and integration of reward and alterations in this system have been observed in addicted populations. Specifically, 1) striatal dopamine is released in response to rewarding substances and experiences, 2) striatal dopamine2/3 receptor densities are lower in cocaine, alcohol, opioid, and nicotine dependent, as well as obese, subjects, and 3) reward-induced striatal dopamine efflux has been shown to be decreased in addicted, relative to non-addicted, subjects.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 21-40
* Tan at least twice weekly over the last year (Frequent Tanners)
* Tan less than twice a week over the last year (Infrequent Tanners)
* Meet modified DSM-IV criteria for Frequent Tanners

Exclusion Criteria:

* Medications that effect brain functioning
* Other medical or psychiatric disorders that may affect neural functioning.
* Drug and Alcohol abuse or dependence
* Pregnancy

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited though flyers and advertisements. Advertisements will be placed in college newspapers. Flyers will be placed on college campuses, and local Dallas stores and beauty salons.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Striatal dopaminergic efflux | Up to one hour post-administration of UVR
  Determine if UVR induces striatal dopaminergic efflux is altered in compulsive tanners.

SECONDARY OUTCOMES:
Striatal D2 receptors | 90 minutes prior to UVR administration
  Basal striatal D2 receptors will be assessed in infrequent and compulsive tanners.

CONTACTS AND LOCATIONS:
Overall Officials: Bryon Adinoff, M.D., Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Division on Addictions, Dallas, Texas, United States

REFERENCES:
- See also: Related Info — http://ais.swmed.edu/redcap/surveys/?s=IJsQqx